CLINICAL TRIAL: NCT04986111
Title: The Efficacy of Purse-string Skin Closure With Negative Pressure Wound Therapy (NPWT) on Wound Recovery After Ileostomy Reversal: A Prospective Randomized Clinical Trial
Brief Title: The Efficacy of Purse-string Skin Closure With Negative Pressure Wound Therapy (NPWT) After Ileostomy Reversal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2007/627-003
Record Dates: First submitted 2021-07-13; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Surgical Site Infection; Wound Heal
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear skin closure with wound drain (Experimental): Reduce fluid collection and dead space by inserting drain into the subcutaneous layer using the wound closure method previously used in the experimental center. The linear suture has a relatively quick time to stitch out.
  Interventions: Procedure: Linear skin closure with wound drain
- Purse-string skin closure with negative pressure wound therapy (Active Comparator): Close the wound with a purse-string suture which is better in terms of surgical site infection but known to take a long time for wound healing, and use negative pressure wound therapy to help granulation of tissues and help healing.
  Interventions: Procedure: Purse-string skin closure with negative pressure wound therapy

INTERVENTIONS:
Procedure: Linear skin closure with wound drain — An oval incision is made around the ileostomy and the continuity of the intestinal tract is restored after adhesion division.
  Methods of anastomosis include either side-to-side or end-to-end, hand-sewing or stapling.
  Linear suture of the rectus abdominis fascia layer by layer. A Jackson-Pratt drainage tube is placed in the subcutaneous tissue and vertical mattress suture is performed with a non-absorbable thread.
  Arms: Linear skin closure with wound drain
Procedure: Purse-string skin closure with negative pressure wound therapy — Recover the intestinal continuity after adhesion division by making a circular incision along the ileostomy Methods of anastomosis include either side-to-side or end-to-end, hand-sewing or stapling.
  Linear suture of the rectus abdominis fascia layer by layer. Negative pressure wound therapy is performed after suturing the subcutaneous tissue using absorbable thread.
  Arms: Purse-string skin closure with negative pressure wound therapy

SUMMARY:
Evaluating the effectiveness of the existing 'linear suture + wound drain placement' and 'purse-string suture + negative pressure wound therapy' through a prospective comparative study

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing ileostomy repair at multicenter

Exclusion Criteria:

* Active bacterial infection needing antibiotics before surgery
* parastomal infection before surgery
* uncontrolled diabetes mellitus
* Emergency repair of stoma (ex. stoma prolapse, high output stoma etc...)
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Unsuccessful wound recovery rate | Check at postoperative 30th day and report through study completion, an average of 1 year
  (patients with unsuccessful wound recovery / all enrolled patients) x 100
  **Unsuccessful wound recovery definition: 1) Occurrence of Surgical Site Infection (SSI) or 2) reoperation due to wound complication or 3) delayed healing over 30 days or 4) Out patient department follow up more than 5 times

CONTACTS AND LOCATIONS:
Overall Officials: Duck-Woo Kim, MD PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea